CLINICAL TRIAL: NCT06743698
Title: A Mixed Methods Process Evaluation of a Randomised Controlled Trial (META Trial) to Evaluate the Use of Metformin in HIV-Positive Persons With Pre-Diabetes
Brief Title: META Trial - a Mixed Methods Process Evaluation
Acronym: META
Status: Not yet recruiting | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: University College London Institute for Global Health (Unknown); National Institute for Medical Research, Tanzania (Other Government); Shree Hindu Mandal Hospital, Tanzania (Unknown); Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Other Study IDs: 101145764; ISRCTN77382043 (Other: International Standard Randomised Controlled Trial Number (ISRCTN))
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-12

CONDITIONS: HIV; Pre-diabetes
Keywords: Qualitative Research; Process evaluation; Metformin; Africa; HIV; Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients that participated in the META trial.
- Healthcare staff: Healthcare staff that were involved in the META trial.

SUMMARY:
The aim of this study is to conduct a mixed methods process evaluation of the META trial. Semi-structured interviews, focus groups, and brief questionnaires will be conducted with a purposive sample of participants (patients and healthcare providers) who were involved in the trial to explore the feasibility, acceptability and perceived effectiveness of the trial intervention.

DETAILED DESCRIPTION:
The META trial was a phase II randomised double-blind placebo-controlled trial that is being conducted in Dar es Salaam, Tanzania to evaluate the use of metformin in HIV-positive persons on antiretroviral therapy (ART) with pre-diabetes.

This study aims to explore the feasibility, acceptability and perceived effectiveness of the META trial intervention by conducting qualitative interviews, focus groups, and brief questionnaires with a purposive sample of participants (patients and healthcare providers) in Tanzania who are involved in the META trial.

Data collection will commence during June-July 2025 with a purposive sample of patients and health care professionals who were involved in the trial (n=50-60).

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in the META Trial
* Participants who have the capacity to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants that took part in the META trial will be able to participate in this study. Not all participants involved in the META trial will be included in this study. However, participants will be purposefully sampled to be reflective of the population who participated in the META trial.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Qualitative interview, focus group, and brief questionnaire findings | 8 weeks
  The primary outcome will the findings of in-depth semi-structured qualitative interviews, focus groups, and brief questionnaires with a purposive sample of patients and HCPs who participated in the META trial (n=50-60).

CONTACTS AND LOCATIONS:
Overall Officials: Walter Cullen, MD, Principal Investigator — UCD NUI: University College Dublin

IPD SHARING:
Plan to Share IPD: No
The study data is likely to include details that would render participants' identifiable and therefore cannot be shared publicly.

REFERENCES:
- [Background] Garrib A, Kivuyo S, Bates K, Ramaiya K, Wang D, Majaliwa E, Simbauranga R, Charles G, van Widenfelt E, Luo H, Alam U, Nyirenda MJ, Jaffar S, Mfinanga S; META trial team. Metformin for the prevention of diabetes among people with HIV and either impaired fasting glucose or impaired glucose tolerance (prediabetes) in Tanzania: a Phase II randomised placebo-controlled trial. Diabetologia. 2023 Oct;66(10):1882-1896. doi: 10.1007/s00125-023-05968-7. Epub 2023 Jul 18. PMID 37460828
- See also: What is The META Trial? (webpage) — https://www.inteafrica.org/related-projects/meta-trial/
- See also: Metformin treatment in Africa (META) (webpage) — https://www.ucl.ac.uk/global-health/research/z-research/respond-africa/metformin-treatment-africa-meta